CLINICAL TRIAL: NCT06613945
Title: Endoscopic Retrograde Cholangiopancreatography With and Without Endoscopic Ultrasound Guided Hepaticogastrostomy for Bilateral Biliary Decompression in Malignant Hilar Biliary Obstruction
Brief Title: ERCP With and Without EUS Guided HGS for Bilateral Biliary Decompression in Malignant Hilar Biliary Obstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD.24.08.881
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Malignant Hilar Stricture
Keywords: Malignant Hilar Biliary Obstruction; Endoscopic Retrograde Cholangiopancreatography; Endoscopic Ultrasound Guided Hepaticogastrostomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined EUS-HGS and ERCP biliary drainage (Active Comparator): unilateral metallic stent will be inserted on right side through ERCP and a hepaticogastrostomy transmural stent will be inserted on left side by EUS to secure biliary drainage
  Interventions: Procedure: Combined ERCP and EUS-HGS biliary drainage
- ERCP biliary drainage (Active Comparator): bilateral metallic stents insertion will be attempted through ERCP to secure biliary drainage
  Interventions: Procedure: ERCP biliary drainage

INTERVENTIONS:
Procedure: ERCP biliary drainage — bilateral metallic stents insertion will be attempted through ERCP to secure biliary drainage
  Arms: ERCP biliary drainage
Procedure: Combined ERCP and EUS-HGS biliary drainage — unilateral metallic stent will be inserted on right side by ERCP and a hepaticogastrostomy transmural stent will be inserted on left side by EUS to secure biliary drainage.
  Arms: Combined EUS-HGS and ERCP biliary drainage

SUMMARY:
A prospective randomized clinical trial to evaluate efficacy and safety of combined EUS-HGS and ERCP compared to ERCP for bilateral biliary decompression in advanced malignant hilar biliary obstruction. The primary outcome will be technical success, clinical success, procedural duration, and re-interventions. Secondary outcomes will be the rate of adverse events. patients will be followed up at 1 and 3 month intervals

DETAILED DESCRIPTION:
Bilateral stenting by Endoscopic Retrograde Cholangiopancreatography in malignant hilar biliary obstructions (MHBO) is challenging and technically difficult. EUS hepaticogastrostomy (EUS-HGS) has been increasingly used as an alternative method to achieve internal biliary drainage in MHBO. Because of the difficulty of ERCP in such scenario, the combination of EUS-HGS and ERCP provides a possible chance of longer stent patency with less event of stent clogging Aim of the work: to evaluate efficacy and safety of combined EUS-HGS and ERCP compared to ERCP for bilateral biliary decompression in advanced MHBO.

The inclusion criteria will be presence of inoperable MHBO with elevated liver tests with serum bilirubin at least 3 times above the upper limit of normal The study patients will be randomized in 1:1 ratio to: ERCP biliary drainage (ERCP-BD) group: bilateral metallic stents insertion will be attempted by transpapilary approach. Combined ERCP and EUS-HGS group: unilateral metallic stent will be inserted on right side by transpapilary approach and a transmural stent will be inserted on left side by EUS.

technical success, clinical success, procedural duration, and re-interventions and adverse events will be assesed

ELIGIBILITY:
Inclusion Criteria:

* Presence of inoperable malignant hilar biliary obstruction on magnetic resonance cholangiography, computed tomography and/or direct cholangiography bismuth type III & IV only.
* Histologically confirmed malignant hilar biliary obstruction.
* Elevated serum bilirubin at least 3 times above the upper limit of normal (1.2 mg/dL).
* Absence of duodenal narrowing/obstruction.
* Accept sharing in the study

Exclusion Criteria:

* Pregnancy.
* Distal biliary obstruction as the main lesion.
* Benign biliary stenosis.
* Malignant hilar biliary obstruction bismuth type I and II.
* Presence of duodenal obstruction.
* Surgically altered anatomy or inability to access the major duodenal papilla.
* Patients underwent previous intervention for biliary drainage.
* Previously failed biliary cannulation at ERCP.
* Large volume ascites.
* Patients unfit for anesthesia.
* Patients having uncorrectable coagulopathy or thrombocytopenia.
* History of allergy to radiocontrast agents.
* Refuse sharing in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Technical success | during the procedure
  considered after stent placement (expanded and patent) with good bile flow and drainage
Procedural duration | at the end of the procedure
  defined as time from biliary cannulation to stent placement by ERCP, and time from needle puncture of the dilated bile duct to stent placement by EUS
Clinical success | 3 month
  considered at 2 weeks by a 50% decrease in total bilirubin levels from baseline and at 4 weeks if total bilirubin is less than 3mg/dL.
Re-interventions | 3 month
  need for re-intervention to secure biliary drainage

SECONDARY OUTCOMES:
Adverse events | 3 month
  Early adverse events (within 48 hours after procedure) including: pancreatitis, cholangitis, bleeding, perforation and peritonitis.
  - Late adverse events include stent dysfunction either due to food impaction, tumor ingrowth or stent migration

CONTACTS AND LOCATIONS:
Overall Officials: Mennatallah E saad, asslecturer, Principal Investigator — Mansoura University
Locations (1):
- Mansoura univeristy, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
the study just started recuriting and the decision to share will be decided when we have prelaminary satisfactory results